CLINICAL TRIAL: NCT06383585
Title: Evaluation of 3D DL oZTEo in the Detection of Osseous Changes in Patients With Inflammatory Arthritis
Brief Title: 3D DL Ozteo in the Detection of Osseous Changes in Patients With Inflammatory Arthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Naveen S. Murthy, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24-001367
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Inflammatory Arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- oZTEo MRI pulse sequence (Experimental): All patients will have the FDA approved MRI pulse sequence, oZTEo, added to their already ordered standard of care MRI examination.
  Interventions: Device: oZTEo

INTERVENTIONS:
Device: oZTEo — An FDA approved MRI pulse sequence, oZTEo, will be added to a standard of care MRI examination. The oZTEo pulse sequence will be anonymized and sent to GE Healthcare for the application of a deep learning algorithm, 3D DL.
  Other Names: 3D DL oZTEo

SUMMARY:
This project intends to explore and validate the utility of new MRI pulse sequence, 3D DL oZTEo, in the detection of osseous erosions of the hand in patients with inflammatory arthritis. The detection of osseous structural changes, such as erosive disease, is routinely assessed in patients with rheumatic conditions such as rheumatoid arthritis, as it alters clinical management, and in some cases assists in diagnosis. Currently, this is most often assessed with radiography and conventional MRI.

DETAILED DESCRIPTION:
This project intends to explore and validate the utility of new MRI pulse sequence, 3D DL oZTEo, in the detection of osseous erosions of the hand in patients with inflammatory arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥18 years of age
* Hand radiographs performed within the past 3-6 months with imaging results available for analysis
* Hand radiographs confirm the presence of bony erosions
* Scheduled for a hand MRI as part of their routine clinical care at Mayo Clinic Rochester

Exclusion Criteria:

- Less than18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The binary (yes/no) presence of bony erosions as detected by hand MRI with and without the addition of the 3D DL oZTEo sequence. | 1 day
  The primary outcome

SECONDARY OUTCOMES:
The number of erosions (continuous) as detected by hand MRI with and without the addition of the 3D DL oZTEo sequence. | 1 day
  The secondary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Naveen Murthy, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials